CLINICAL TRIAL: NCT02447718
Title: Vaccinating Children After Chemotherapy for Acute Lymphoblastic Leukemia: A Canadian Immunization Research Network Study
Brief Title: Vaccinating Children After Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Responsible Party: Principal Investigator, Karina Top, Principal Investigator, Canadian Immunization Research Network
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SI02
Record Dates: First submitted 2015-05-13; First posted 2015-05-19 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Active Comparator): Children who were diagnosed with ALL at ≥1 year of age, and are within 6-8 months of completing chemotherapy will receive 1 dose each of: Prevnar®13 and Pediacel® vaccines, followed by 1 dose of Pneumovax® 23 given 2 months after PCV13.
  Interventions: Biological: Prevnar®13; Biological: Pneumovax® 23; Biological: Pediacel®
- Healthy Control (No Intervention): Children 3-18 years of age who are not immunocompromised age-matched to cases from Group 1.

INTERVENTIONS:
Biological: Prevnar®13 — A single dose of Prevnar®13 will be administered to subjects with ALL who are 6-12 months post-completion of chemotherapy.
  Other Names: 13- valent conjugate pneumococcal vaccine; PCV13
  Arms: Experimental
Biological: Pneumovax® 23 — A single dose of Pneumovax® 23 will be administered to subjects approximately 2 months after Prevnar®13
  Other Names: 23-valent polysaccharide pneumococcal vaccine; PPV23
  Arms: Experimental
Biological: Pediacel® — A single dose of Pediacel® will be administered to subjects with ALL who are 6-12 months post-completion of chemotherapy.
  Other Names: DTaP-IPV-Hib
  Arms: Experimental

SUMMARY:
This multi-center open label clinical trial aims to identify predictors of low antibody titers to vaccine antigens in children with ALL who completed chemotherapy in the prior 6 months, and to determine the immunogenicity and safety of diphtheria-tetanus-acellular pertussis-inactivated poliomyelitis-Haemophilus influenzae type b (DTaP-IPV-Hib) and 13-valent pneumococcal conjugate vaccine (PCV13) booster immunization administered 6 months post-chemotherapy, followed by 23-valent pneumococcal polysaccharide vaccination (PPV23) 2 months later. The results will support the development of clinical practice guidelines for this population.

DETAILED DESCRIPTION:
Rationale and Aims: Children with acute lymphoblastic leukemia (ALL) have evidence of persistent immunosuppression following chemotherapy and may experience waning of immunity to vaccines received prior to treatment. There is no standard of care in Canada regarding immunologic evaluation or booster immunization of children with ALL after chemotherapy. This study aims to identify predictors of low baseline immunity to vaccine antigens in children with ALL and to evaluate the immunogenicity and safety of a standard immunization regimen: DTaP-IPV-Hib and PCV13 booster immunization administered 6 months post-chemotherapy, followed by PPV23.

Study Design: This will be a multi-center open-label clinical trial in which children who were diagnosed with ALL at ≥1 year of age, and have not received immunizations other than influenza since completing chemotherapy will undergo immunologic evaluation and serologic testing for pneumococcus, tetanus, pertussis and varicella. They will then be immunized with PCV13, DTaP-IPV-Hib, regardless of immunization history [unless PPV23 was received within the prior 12 months]. Other routine vaccines required as per provincial and centre-specific immunization policies will also be administered. PPV23 will be administered 8 weeks after PCV13. Repeat serologic testing will be conducted at 2 months and 12-15 months after DTaP-IPV-Hib and PCV13 immunization to assess short and long-term immune responses.

Adverse events following immunization (AEFI) will be captured through standardized telephone interviews on days 8-10 and 30-33 post-immunization that will capture local and systemic AEFI.

ELIGIBILITY:
Cases with ALL:

Inclusion Criteria:

* Diagnosed with standard, high-risk or very-high risk ALL
* Age at diagnosis: ≥1 year of age (age at enrollment: ≥3 years)
* Completed chemotherapy 3 to 12 months prior to enrollment
* No evidence of ALL relapse or secondary malignancy
* No known primary immunodeficiency
* No receipt of pneumococcal or tetanus-containing vaccines since completing chemotherapy
* No history of allergy to any component of PCV13
* Caregiver and/or participant is English or French-speaking and able to provide written informed consent

Exclusion Criteria:

* Infantile ALL
* Evidence of disease relapse or secondary malignancy
* History of underlying primary immunodeficiency
* Transplant recipient
* Received intravenous immunoglobulin (IVIG) within past 9 months or other blood products within the prior 3 months.Children who received PPV23 within 12 months of enrollment will not be eligible to receive PCV13 or PPV23. These children can still participate in the baseline evaluation, receive DTaP-Hib-IPV vaccine, and have tetanus and pertussis serology measured at 2 and 12-15 months post-immunization.

Controls:

Inclusion criteria

* Children 3-18 years of age, age-matched to cases
* Caregiver and/or participant is English or French-speaking and able to provide written informed consent

Exclusion criteria

* History of primary or secondary immunodeficiency including aplastic anemia, malignancy, nephrotic syndrome, malabsorption or severe malnutrition
* Immunosuppressive therapy within 3 months of enrollment (excluding inhaled corticosteroids)
* Received intravenous immunoglobulin (IVIG) within past 9 months or other blood products within the prior 3 months.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Top, MD, MS, Principal Investigator — Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Top KA, Vaudry W, Morris SK, Pham-Huy A, Pernica JM, Tapiero B, Gantt S, Price VE, Rassekh SR, Sung L, McConnell A, Rubin E, Chawla R, Halperin SA. Waning Vaccine Immunity and Vaccination Responses in Children Treated for Acute Lymphoblastic Leukemia: A Canadian Immunization Research Network Study. Clin Infect Dis. 2020 Dec 3;71(9):e439-e448. doi: 10.1093/cid/ciaa163. PMID 32067048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral across 10 pediatric centres. Controls were recruited at 3 centres. Participants were enrolled between November 2015 to September 2017.
Pre-assignment Details: 155 of the 156 participants recruited met inclusion criteria. Of the 78 participants with ALL recruited, 1 did not meet inclusion criteria and 3 withdrew consent prior to study start. All of the 78 control participants met inclusion criteria.
Period: Overall Study
Arm/Group | Experimental | Healthy Control
Started | 78 | 78
Received Prevnar®13 | 74 | 0 (Do not receive vaccination)
Received Pediacel® | 73 | 0 (Do not receive vaccination)
Received Pneumovax® 23 | 73 | 0 (Do not receive vaccination)
Completed | 66 | 78
Not Completed | 12 | 0
Not completed — Lost to Follow-up | 8 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Screen Failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Healthy Control | Total
Number analyzed (Participants) | 74 | 78 | 152
Age, Continuous [Mean (Full Range); unit: years] | 8.1 [3.8 to 19.3] | 8.3 [3.5 to 18.9] | 8.2 [3.5 to 19.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 37 | 40 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 74 | 78 | 152
ALL disease risk category [Count of Participants; unit: Participants] — Disease risk category based on patient characteristics at leukemia diagnosis reflects intensity of chemotherapy Population: Only collected for ALL participants
  Participants
    Standard risk: number analyzed (Participants) | 74 | 0 | 74
    Standard risk | 40 |  | 40
    High risk: number analyzed (Participants) | 74 | 0 | 74
    High risk | 27 |  | 27
    Very high risk: number analyzed (Participants) | 74 | 0 | 74
    Very high risk | 6 |  | 6
    Unknown: number analyzed (Participants) | 74 | 0 | 74
    Unknown | 1 |  | 1
Treatment Protocol [Count of Participants; unit: Participants] — Population: Only collected for ALL participants
  Participants
    Children's Oncology Group: number analyzed (Participants) | 74 | 0 | 74
    Children's Oncology Group | 49 |  | 49
    Dana Farber Cancer Institute: number analyzed (Participants) | 74 | 0 | 74
    Dana Farber Cancer Institute | 25 |  | 25
Interval from last chemotherapy to serology [Median (Full Range); unit: months] — Time in months between last chemotherapy session to baseline blood draw. Population: Only collected for ALL participants
  months
    number analyzed (Participants) | 74 | 0 | 74
    (all) | 6 [4 to 10] |  | 6 [4 to 10]
Total white blood cell count at enrollment [Median (Inter-Quartile Range); unit: cells x10^9/l] — Only available for participants with analyzable data Population: Only collected for participants with AL. Immunological markers not available on all participants with ALL, denominator reflects number of participants with analyzable values for each test.
  cells x10^9/l
    number analyzed (Participants) | 69 | 0 | 69
    (all) | 6.5 [5.3 to 7.7] |  | 6.5 [5.3 to 7.7]
Total lymphocyte count at enrollment [Median (Inter-Quartile Range); unit: cells x10^9/l] — Only available for participants with analyzable data Population: Only collected for participants with ALL. Immunological markers not available on all participants with ALL, denominator reflects number of participants with analyzable values for each test.
  cells x10^9/l
    number analyzed (Participants) | 73 | 0 | 73
    (all) | 2.3 [1.7 to 2.9] |  | 2.3 [1.7 to 2.9]
Lymphocyte subsets at enrollment [Median (Inter-Quartile Range); unit: cells x10^9/l] — Population: Only collected for participants with ALL. Immunological markers not available on all participants with ALL, denominator reflects number of participants with analyzable values for each test.
  cells x10^9/l
    CD3+ T cells: number analyzed (Participants) | 60 | 0 | 60
    CD3+ T cells | 1.4 [1.1 to 1.9] |  | 1.4 [1.1 to 1.9]
    CD4+ T cells: number analyzed (Participants) | 60 | 0 | 60
    CD4+ T cells | 0.8 [0.6 to 1.0] |  | 0.8 [0.6 to 1.0]
    CD8+ T cells: number analyzed (Participants) | 60 | 0 | 60
    CD8+ T cells | 0.5 [0.3 to 0.7] |  | 0.5 [0.3 to 0.7]
    NK cells (CD56+/CD16+): number analyzed (Participants) | 60 | 0 | 60
    NK cells (CD56+/CD16+) | 0.2 [0.1 to 0.2] |  | 0.2 [0.1 to 0.2]
    CD19+ B cells: number analyzed (Participants) | 60 | 0 | 60
    CD19+ B cells | 0.6 [0.4 to 0.7] |  | 0.6 [0.4 to 0.7]
Total serum IgG at enrollment [Median (Inter-Quartile Range); unit: g/l] — Only available for participants with analyzable data Population: Only collected for participants with ALL. Immunological markers not available on all participants with ALL, denominator reflects number of participants with analyzable values for each test.
  g/l
    number analyzed (Participants) | 71 | 0 | 71
    (all) | 8.5 [7.1 to 11.1] |  | 8.5 [7.1 to 11.1]
Previous doses of PCV [Count of Participants; unit: Participants]
  0 | 19 | 9 | 28
  1-2 | 10 | 2 | 12
  ≥3 | 45 | 66 | 111
  Unknown | 0 | 1 | 1
  Received more than ≥1 dose at ≥12 months of age | 44 | 62 | 106
  Received more than ≥1 dose PCV13 | 34 | 38 | 72
Previous doses of DTaP or Tdap [Count of Participants; unit: Participants]
  0 | 2 | 0 | 2
  1-3 | 12 | 1 | 13
  4 | 36 | 17 | 53
  ≥5 | 24 | 60 | 84
Previous doses of varicella vaccine [Count of Participants; unit: Participants]
  0 | 17 | 11 | 28
  1 | 48 | 26 | 74
  ≥2 | 9 | 40 | 49
  Unknown | 0 | 1 | 1
Interval from last vaccine to baseline blood draw [Mean (Standard Deviation); unit: years]
  DTaP/Tdap-containing vaccine | 6.0 (2.7) | 3.7 (2.5) | 4.85 (2.6)
  PCV | 5.4 (2.3) | 7.2 (3.4) | 6.3 (2.85)
  Varicella | 6.5 (3.2) | 5.2 (4.2) | 5.85 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Protective Titres to PCV13 Serotypes Post-immunization With PCV13+PPV23
Description: The percentage of participants with protective titres (with protective level defined as ≥0.35 ug/ml, as per World Health Organization criteria) to PCV13 serotypes will be assessed at 2 months and 12-15 months post PCV13+PPV23 and compared to baseline levels.
Time Frame: Pre-vaccination Baseline, 2 months and 12-15 months
Population: Participants analyzed equaled the overall number of ALL participants that completed the study and had analyzable serology collected at 2 months and 12-15 months post-vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 66
Participants
  2 months post-PCV13 | 40
  12-15 months post-PCV13 | 22

2. Secondary Outcome: Number of Participants With Protective Titres to PCV7 Serotypes at Baseline
Description: The number of participants with protective titres (≥0.35 ug/ml) to PCV7 serotypes at baseline will be compared to age-matched controls.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Healthy Control
Number analyzed (Participants) | 73 | 78
Participants | 4 | 30

3. Secondary Outcome: Baseline Pneumococcal Antibody Titres in Subjects With ALL Versus Controls
Description: Baseline geometric mean titers (GMT) and percentage of subjects with protective titres to pneumococcal serotypes in children with ALL versus age-matched controls.
Time Frame: Day 0
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Experimental | Healthy Control
Number analyzed (Participants) | 73 | 78
mg/L
  Pneumococcal Serotype 1 | 0.19 [0.16 to 0.22] | 0.52 [0.41 to 0.66]
  Pneumococcal Serotype 3 | 0.17 [0.14 to 0.21] | 1.01 [0.72 to 1.42]
  Pneumococcal Serotype 4 | 0.19 [0.16 to 0.22] | 0.54 [0.43 to 0.68]
  Pneumococcal Serotype 6B | 0.38 [0.29 to 0.50] | 1.20 [0.92 to 1.57]
  Pneumococcal Serotype 7F | 0.26 [0.20 to 0.33] | 0.7 [0.57 to 0.87]
  Pneumococcal Serotype 9V | 0.45 [0.37 to 0.55] | 0.92 [0.77 to 1.10]
  Pneumococcal Serotype 14 | 0.46 [0.35 to 0.59] | 1.76 [1.24 to 2.50]
  Pneumococcal Serotype 18C | 0.21 [0.16 to 0.27] | 0.49 [0.38 to 0.62]
  Pneumococcal Serotype 19F | 0.99 [0.77 to 1.26] | 3.21 [2.73 to 3.76]
  Pneumococcal Serotype 23F | 0.29 [0.23 to 0.36] | 1.15 [0.87 to 1.52]

4. Secondary Outcome: Immune Responses to Pertussis Toxin Following DTaP-IPV-Hib Booster Vaccination
Description: Baseline, Short-term (baseline - 2 months after vaccination) and long-term (baseline - 12-15 months) vaccine responses to DTaP-IPV-Hib will be measured using GMT ratios.
Time Frame: Prevaccination baseline, 2 months, 12-15 months
Population: A total of 73 participants received DTaP-IPV-Hib, 67 provided a follow up sample at 2 months post-vaccination and 66 provided a follow up sample at 12 months post-vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/ml
Groups:
- Experimental: Children who were diagnosed with ALL at ≥1 year of age, and are within 6-8 months of completing chemotherapy will receive 1 dose each of: Prevnar®13 and Pediacel® vaccines, followed by 1 dose of Pneumovax® 23 given 2 months after PCV13.
  Prevnar®13: A single dose of Prevnar®13 will be administered to subjects with ALL who are 6-12 months post-completion of chemotherapy.
  Pneumovax® 23: A single dose of Pneumovax® 23 will be administered to subjects approximately 2 months after Prevnar®13 Pediacel®: A single dose of Pediacel® will be administered to subjects with ALL who are 6-12 months post-completion of chemotherapy.
Arm/Group | Experimental
Number analyzed (Participants) | 73
EU/ml
  Pre-vaccination Baseline | 4.10 [3.67 to 4.58]
  Baseline - 2 months post-vaccination: number analyzed (Participants) | 67
  Baseline - 2 months post-vaccination | 30.67 [22.25 to 42.29]
  Baseline - 12-15 months post-vaccination: number analyzed (Participants) | 66
  Baseline - 12-15 months post-vaccination | 10.39 [7.76 to 13.91]

5. Secondary Outcome: Baseline Tetanus Toxoid Antibody Titers in Children With ALL Versus Controls
Description: Baseline geometric mean titers (95% confidence intervals) reported as IU/ml in children with ALL versus controls
Time Frame: Day 0
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Experimental | Healthy Control
Number analyzed (Participants) | 73 | 78
IU/ml | 0.16 [0.12 to 0.20] | 1.73 [1.26 to 2.37]

6. Secondary Outcome: Baseline Pertussis Toxin Titers in Children With ALL Versus Healthy Controls
Description: Baseline geometric mean titers (95% confidence intervals) reported as IU/ml in children with ALL versus controls
Time Frame: Day 0
Measure: Geometric Mean (95% Confidence Interval); unit: EU/ml
Arm/Group | Experimental | Healthy Control
Number analyzed (Participants) | 73 | 78
EU/ml | 4.10 [3.67 to 4.58] | 10.35 [8.15 to 13.16]

7. Secondary Outcome: Baseline Varicella Titers in Children With ALL Versus Controls.
Description: Geometric mean titers (95% confidence interval) in AI (antibody index)
Time Frame: Day 0
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody index
Arm/Group | Experimental | Healthy Control
Number analyzed (Participants) | 73 | 78
Antibody index | 0.33 [0.24 to 0.45] | 1.00 [0.77 to 1.29]

8. Secondary Outcome: Immune Responses to Tetanus Toxoid Following DTaP-IPV-Hib Immunization
Description: Baseline, short-term (baseline to 2 months after vaccination) and long-term (baseline to 12-15 months) vaccine responses to DTaP-IPV-Hib will be measured using GMTs with 95% confidence intervals
Time Frame: baseline, 2 months, 12-15 months
Population: Participants with analyzable data at each timepoint were included
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Experimental
Number analyzed (Participants) | 73
IU/ml
  Pre-vaccination Baseline | 0.16 [0.12 to 0.20]
  Baseline - 2 months post-vaccination | 4.00 [2.57 to 6.22]
  Baseline - 12-15 months post-vaccination | 1.08 [0.77 to 1.52]

9. Other Pre Specified Outcome: Number of Participants With Adverse Events Following Immunization Requiring Healthcare Visit or Leading to >=1 Day of Disability
Description: Adverse Events Following Immunization requiring healthcare visit or leading to >=1 day of disability will be captured through structured telephone interviews on days 8-10 and 30-33 after each immunization
Time Frame: days 8-10 and 30-33
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 74
Participants
  Possibly related to vaccination | 3
  Unrelated to vaccination | 7
  No AEFI requiring healthcare visit or leading to >=1 day of disability | 64

ADVERSE EVENTS:
Time Frame: AEFI was captured through structured telephone interviews on days 8-10 and 30-33 after each immunization
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse Events were not monitored for Healthy Controls as they did not receive the interventions, they provided baseline data only.
Groups:
- DTaP-IPV-HiB+PCV13: DTaP-IPV-Hib: diphtheria-tetanus-acellular pertussis-inactivated polio-H. influenzae type b vaccine
  PCV13: 13-valent pneumococcal conjugate vaccine
- PPV23: PPV23: 23-valent pneumococcal polysaccharide vaccine
Arm/Group | DTaP-IPV-HiB+PCV13 | PPV23
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/73
Other Adverse Events (participants affected / at risk) | 56/74 | 46/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTaP-IPV-HiB+PCV13 (N=74) | PPV23 (N=73)
Pain/erythema/swelling at injection site (Skin and subcutaneous tissue disorders) | 52 | 45
Systemic symptoms (General disorders) | 18 | 12 — Systemic symptoms included fever, malaise, gastrointestinal symptoms, skin rash, headache, pharyngitis, otitis media

LIMITATIONS AND CAVEATS:
1. Antibody levels to vaccine antigens were not measured before chemotherapy, cannot confirm that chemotherapy was the cause of low postchemotherapy titers.
2. Immunization status at ALL diagnosis was not assessed and therefore could not confirm whether postchemotherapy participants were underimmunized for age before diagnosis relative to their peers.
3. We were unable to assess antibodies to other pertussis antigens (eg, filamentous hemagglutinin, pertactin), only anti-PT antibodies alone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT02447718/Prot_SAP_000.pdf